CLINICAL TRIAL: NCT04331522
Title: Allergen Provocations at Hans Christian Andersen Children's Hospital
Brief Title: Allergen Provocations- HCA Children's Hospital
Status: Recruiting | Type: Observational
Sponsor: Josefine Gradman (Other)
Responsible Party: Sponsor-Investigator, Josefine Gradman, Consultant, phd, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: HCA-AP
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Allergy in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 17 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (15):
- Antibiotics: Children aged 0-18 years investigated for allergy to antibiotics
  Interventions: Diagnostic Test: Oral provocation test
- Milk: Children aged 0-18 years investigated for allergy to milk
  Interventions: Diagnostic Test: Oral provocation test
- Egg: Children aged 0-18 years investigated for allergy to egg
  Interventions: Diagnostic Test: Oral provocation test
- Peanut: Children aged 0-18 years investigated for allergy to peanut
  Interventions: Diagnostic Test: Oral provocation test
- Hazelnut: Children aged 0-18 years investigated for allergy to hazelnut
  Interventions: Diagnostic Test: Oral provocation test
- Sesame: Children aged 0-18 years investigated for allergy to sesame
  Interventions: Diagnostic Test: Oral provocation test
- Wheat: Children aged 0-18 years investigated for allergy to wheat
  Interventions: Diagnostic Test: Oral provocation test
- walnut: Children aged 0-18 years investigated for allergy to walnut
  Interventions: Diagnostic Test: Oral provocation test
- cashew: Children aged 0-18 years investigated for allergy to cashew
  Interventions: Diagnostic Test: Oral provocation test
- Pistachio: Children aged 0-18 years investigated for allergy to pistachio
  Interventions: Diagnostic Test: Oral provocation test
- Almond: Children aged 0-18 years investigated for allergy to almond
  Interventions: Diagnostic Test: Oral provocation test
- Soy: Children aged 0-18 years investigated for allergy to soy
  Interventions: Diagnostic Test: Oral provocation test
- Fish: Children aged 0-18 years investigated for allergy to fish
  Interventions: Diagnostic Test: Oral provocation test
- Shellfish: Children aged 0-18 years investigated for allergy to shellfish
  Interventions: Diagnostic Test: Oral provocation test
- Poppy seed: Children aged 0-18 years investigated for allergy to poppy seed
  Interventions: Diagnostic Test: Oral provocation test

INTERVENTIONS:
Diagnostic Test: Oral provocation test — Titrated provocation with allergen

SUMMARY:
A prospective study of all allergen provocations performed in children at the Hans Christian Andersen Children's Hospital.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the impact of co-morbidities, history, and allergen tests on the outcome of allergen provocation tests.

Subjects are children aged 0-18 years old investigated for allergy to foods or antibiotics. Data entered in the database are demographics, co-morbidities, symptoms, SPT, specific IgE and details of the allergen provocations.

ELIGIBILITY:
Inclusion Criteria:

clinical suspicion of allergy to foods or antibiotics informed concent -

Exclusion Criteria:

-

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children referred to the department of pediatrics for investigation of allergy to foods or antibiotics
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2038-10 (Estimated); Study Completion 2039-10 (Estimated)

PRIMARY OUTCOMES:
The association of allergy tests with the result of allergen provocation | 5 years
  The value of specific IgE and SPT to predict the outcome of a allergen provocation

CONTACTS AND LOCATIONS:
Locations (1):
- Hans Christian Andersen Children's Hospital, Odense, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gradman J, Petersen BT, Halken S. Oral food challenge with raw egg: Sixty-minute- compared with 30-minute dosing interval. Clin Exp Allergy. 2022 Sep;52(9):1114-1117. doi: 10.1111/cea.14187. Epub 2022 Jul 4. No abstract available. PMID 35719001
- [Derived] Petersen BT, Gradman J. Prospective study of 5-day challenge with penicillins in children. BMJ Paediatr Open. 2020 Aug 4;4(1):e000734. doi: 10.1136/bmjpo-2020-000734. eCollection 2020. PMID 32818157